CLINICAL TRIAL: NCT02566486
Title: Postoperative Pain Intensity After Using Different Instrumentation Techniques: a Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ersan Çiçek, Assistant Professor, PhD, Bulent Ecevit University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-27194235-03
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reciprocating system (Other): Waveone root canal instrumentation file
  Interventions: Device: Reciprocating system
- Rotational system (Other): ProTaper Next root canal instrumentation file
  Interventions: Device: Rotational system

INTERVENTIONS:
Device: Reciprocating system — Different root canal instrumentation systems
  Other Names: WaveOne
  Arms: Reciprocating system
Device: Rotational system — Different root canal instrumentation systems
  Other Names: ProTaper Next
  Arms: Rotational system

SUMMARY:
Aim The aim of this clinical study was to evaluate the influence of the instrumentation techniques on the incidence and intensity of postoperative pain in single-visit root canal treatment.

Methodology Ninety patients with single root/canal and non-vital pulps were included. The patients were assigned into 3 groups according to root canal instrumentation technique used; the modified step-back (stainless-steel hand files, HF), reciprocal (WaveOne, WO), and rotational (ProTaper Next, PTN). Root canal treatment was carried out in a single visit and the severity of postoperative pain was assessed by 4-point pain intensity scale. All the participants were called through phone at 12, 24 and 48 h to obtain the pain scores. Data were analyzed by the Kruskal-Wallis test.

DETAILED DESCRIPTION:
Overall, 90 patients who had asymptomatic and non-vital teeth associated with periapical lesions, were included to the study. All diagnosis and treatment procedures were performed by a single operator to eliminate or minimize individual variability in the treatment between clinicians. The patients were randomly stratified into 3 groups of 30 by coin toss. Allocation was done by a person other than the operator performing the root canal procedure. The patients were assigned into three equal groups according to instrumentation techniques used (n=30);

* The modified step-back technique (n=30): The canals were instrumented with a modified step-back technique using stainless-steel hand files (HF, Dentsply Maillefer, Ballaigues, Switzerland). The canals were prepared to a master apical size 02/40 with K files by using the balance force technique. Step back technique was performed by using K-files #45-55 to a master apical size 02/40 with K files. The step back technique was performed using K-files #45-55.
* Reciprocal technique (n=30): The canals were instrumented with a driven reciprocation motion, using WaveOne (WO, Dentsply Maillefer, Ballaigues, Switzerland) file having a size 40 and a taper of 0.06 slow in-and-out pecking motion according to the manufacturer's instructions. The flutes of the instrument were cleaned after 3 pecks.
* Rotational technique (n=30): The canals were instrumented using ProTaper Next (PTN, Dentsply Maillefer, Ballaigues, Switzerland) 06/40 file in the sequence X1, X2, X3, X4 at a rotational speed of 300 rpm and 200 g/cm torque according to the manufacturer's instructions. The instruments were used up to the working length.

After isolation and access cavity preparation, the initial working length was then determined with an electronic root canal measurement device (Root ZX mini; J. Morita, Tokyo, Japan). It was confirmed using periapical radiographs. During the instrumentation, a total of 10 ml of 5% NaOCl were used for irrigation. The irrigation needle (NaviTip 31ga needle; Ultradent, South Jordan, UT, USA) was placed as deep as possible into the canal without resistance until it was 1 mm short of the predetermined WL.The final irrigation was performed with 5% NaOCl, 17% EDTA, and 2% chlorhexidine.

The root canals were obturated with gutta-percha and a resin based sealer (AH26, De Trey Dentsply, Konstanz, Germany) using cold lateral compaction technique. A standardized master cone size #40.02 gutta-percha was fitted with tug back at the working length. The gutta-percha cone was lightly coated with sealer and slowly inserted into the canal. Cold lateral compaction with accessory gutta-percha cones size 15 was performed until these could not be introduced more than 5 mm into the root canal. All canals were shaped, cleaned, and obturated in a single-visit.

Although no systemic medication was prescribed, the patients were instructed to take mild analgesics (400 mg of ibuprofen), if they experienced pain. The assessment of postoperative pain was carried out at 12, 24, and 48 hours after initial appointment by one independent clinician blinded to the groups. All the participants were called by blinded operator through phone at 12, 24 and 48 h to obtain the pain scores using a 4-point pain intensity scale (Dalton Orstavik et al. 1998). The presence or absence of pain, or the appropriate degree of pain was recorded by using a 4-point pain intensity scale. The pain categories were as follows:

1. no pain;
2. slight pain (mild discomfort, need no treatment);
3. moderate pain (pain relieved by analgesics);
4. severe pain (pain and/or swelling not relieved by simple analgesics and required unscheduled visit).

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic and non-vital teeth associated with periapical lesions

Exclusion Criteria:

* vital tooth

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
4-point pain intensity scale | 48 hours
  Change from intensity of postoperative pain at 48 hours